CLINICAL TRIAL: NCT05074797
Title: Epidemology of Acute Kidney Injury in Diabetic Patients Infected With covid_19 In Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Doaa Rmadan, Doaa011180@med.aun.edu.eg, Assiut University
Other Study IDs: Acute kidney in covid_19
Record Dates: First submitted 2021-10-01; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Acute Kidney Injury Due to covid_19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- covid not diabetic with AKI: AKI in pt with covid_19 not diabetic
  Interventions: Diagnostic Test: laboratory
- AKI in covid_19 in diabetic: AKI in covid_19 in diabetic pt
  Interventions: Diagnostic Test: laboratory
- covid_19 in diabetic: covid_19 in diabetic without AKI
  Interventions: Diagnostic Test: laboratory

INTERVENTIONS:
Diagnostic Test: laboratory — laboratory data

SUMMARY:
The novel coronavirus SARS-CoV-2 was identified as the causative agent for a series of atypical respiratory diseases in Wuhan, China in December of 2019(.1) The disease termed COVID-19, was officially declared a pandemic by the World Health Organization on March 11, 2020. SARS-CoV-2 contains a single-stranded, positive-sense RNA genome surrounded by an extracellular membrane containing a series of spike glycoproteins resembling a crown.COVID-19 infection results in diverse symptoms and morbidity depending on individual genetics, ethnicity, age, and geographic location. In severe cases, COVID-19 pathophysiology includes destruction of lung epithelial cells, thrombosis, hypercoagulation, and vascular leak leading to sepsis.(2) COVID-19 risk factors include cardiovascular disease, hypertension, and diabetes.(2)

DETAILED DESCRIPTION:
Notably, in several studies, diabetes is one of the most reported comorbidities with poor prognosis in patients with severe COVID-19 due to Compromised innate immunity, pro-inflammatory cytokine reduced expression of ACE2 and use of renin-angiotensin-aldosterone system antagonists. (3) On the other hand, COVID-19 contributes to worsening of dysglycemia in people with diabetes mellitus by direct β-cell damage, cytokine-induced insulin resistance, hypokalemia and drugs used in the treatment of COVID-19 (like corticosteroids, lopinavir/ritonavir).(4) Nearly half of critically ill patients would develop AKI at some point during their ICU admission.(5) Acute kidney injury (AKI) has been reported to be the second observed complication in deceased patients after ARDS.it is reported that patients who died with covid19 had different degrees of AKI .The pathogenesis of kidney injury in patients infected with covid19 is multifactorial: (1) prerenal azotemia, ATN can occur owing to many contributing factors including volume depletion, cytokine storm, hypoxia, shock, or rhabdomyolysis (2) proximal tubular injury, (3) glomerulopathy, (4) thrombotic microangiopathy, and (5)complications from the treatment of COVID_19. (6)

ELIGIBILITY:
Inclusion Criteria:

* patients admitted because of COVID-19 infetion.

Exclusion Criteria:

* Patients with ESRD on regular dialysis ,Patients with stage 4 or 5 non-dialysis if the condition proven to be progression of the already known diagnosis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Data will be collected by a questionnaire includes the followings:
  * Socio demographic data (name, age, sex, Body weight and height, job, marital status, number of children, educational level and residence etc).
  * Main presenting symptoms
  * History of hypertension, chronic kidney disease, ect.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-02-20 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
percentage of AKI in covid_19 in diabetic pt | 6 months
  diabetic pt with AKI due to infection with covid _19

CONTACTS AND LOCATIONS:
Overall Officials: doaa DR rezk, master, Principal Investigator — University Hospital
Locations (1):
- Doaa Ramadan Rezk, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided